CLINICAL TRIAL: NCT01760226
Title: Use of Dose Adjusted EPOCH-R in the Treatment of Childhood Mature B Cell Malignancies
Brief Title: Dose Adjusted EPOCH-R, to Treat Mature B Cell Malignancies
Acronym: DA-EPOCH-R
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Carl Allen, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-30759, DA-EPOCH-R; DA-EPOCH-R (Other: BCM); 5K12CA090433-12 (NIH)
Record Dates: First submitted 2012-12-17; First posted 2013-01-04 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2024-02

CONDITIONS: Diffuse Large B Cell Lymphoma; Post Transplant Lymphoproliferative Disorder; Primary Mediastinal (Thymic) Large B-cell Lymphoma
Keywords: DLBCL; Diffuse large B cell lymphoma; dose adjusted; EPOCH; Etoposide; Doxorubicin; Vincristine; Cyclophosphamide; Prednisone; Rituximab
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Methotrexate; Etoposide; Doxorubicin; Vincristine; Rituximab; Cyclophosphamide; Prednisone; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- DA-EPOCH-R for DLBCL, PTLD & PMBCL (Experimental): Minimum of 6 cycles (cycle=3 weeks), possibly 8. Dosages of the drugs will be determined by the subject's weight and height for cycle 1. Thereafter, the dosages of some drugs will be adjusted up or down for the next cycle, dependent on the blood tests results.
  DA-EPOCH-R for 2 cycles then two more cycles of DA-EPOCH-R. If complete response (CR), then DA-EPOCH-R for more 2 cycles. If no CR, DA-EPOCH-R for 4 more cycles.
  Interventions: Drug: DA-EPOCH-R for DLBCL, PTLD, AND PMBCL; Drug: Methotrexate; Drug: Etoposide; Drug: Doxorubicin; Drug: Vincristine; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Prednisone; Drug: G-CSF

INTERVENTIONS:
Drug: DA-EPOCH-R for DLBCL, PTLD, AND PMBCL — Day 1: Rituximab IV
  Days 1-4: After rituximab, etoposide, vincristine, and doxorubicin will be given in a vein over 96 hours as a continuous infusion.
  Day 5: cyclophosphamide will be given in a vein
  Days 1-5: prednisone given by mouth twice a day
  G-CSF 5mcg/kg/day will be given under the skin from day 6 until ANC has improved.
  Other Names: DA-EPOCH-R
Drug: Methotrexate — CNS negative patients with high CNS risk DLBCL will receive age based, intrathecal dosing of MTX on days 1 and 5 of cycles 3 - 6 only.
  CNS positive patients will receive age based, intrathecal (within the spinal fluid) MTX twice weekly for 2 weeks past the first negative cytology with a minimum of 4 weeks treatment. Then, weekly for 6 weeks and then every 4 weeks for 6 months.
  DLBCL/PTLD/PMBCL CNS prophylaxis for cycles 3-6 ONLY if:
  * 2+ extranodal sites
  * elevated LDH,
  * MYC rearrangement OR
  * bone or marrow disease.
  ALL OTHERS receive IT MTX cycles 3-6.
  Other Names: MTX
Drug: Etoposide — Etoposide will be given at 50mg/m2/day on days 1-4 of the first cycle of therapy (dose based on patient height and weight). The doses in later cycles will be adjusted up or down based on the patient's blood test results.
  Other Names: VP-16
Drug: Doxorubicin — Doxorubicin will be given at 10mg/m2/day on days 1-4 of the first cycle (dose based on patient height and weight). The doses in later cycles will be adjusted up or down based on the patient's blood test results.
  Other Names: Adriamycin; hydroxydaunorubicin
Drug: Vincristine — Vincristine will be given on days 1-4 of each cycle at 0.4mg/m2/day (dose based on patient height and weight).
  Other Names: Oncovin; LCR; VCR; Vincasar Pfs
Drug: Rituximab — Rituximab (375mg/m2/dose) will only be given on Day 1 of each cycle prior to all the other chemotherapy agents. Dose is based on patient height and weight.
  Other Names: Rituxan
Drug: Cyclophosphamide — Cyclophosphamide will be given on Day 5 of each cycle. In cycle 1, the dose will be 750 mg/m2 (based on patient height and weight), and the dose will be adjusted up or down for future cycles based on blood test results.
  Other Names: Cytoxan; Neosar; CTX
Drug: Prednisone — Prednisone will be given by mouth at 60mg/m2/dose (based on height and weight) twice a day on days 1-5 of each cycle.
  Other Names: Deltasone
Drug: G-CSF — G-CSF will be given at 5 mcg/kg/day during each cycle, starting on day 6, until the patient's ANC (absolute neutrophil count) is greater than 5000/mcL past nadir.
  Other Names: Neupogen; Granulocyte - Colony Stimulating Factor

SUMMARY:
The subject is invited to take part in this research study because s/he has been diagnosed with Diffuse Large B-Cell Lymphoma (DLBCL), Primary Mediastinal B-cell Lymphoma (PMBCL), or Post-transplant Lymphoproliferative Disorder (PTLD).

In an attempt to improve cure rates while reducing harmful effects from drugs, oncologists are developing new treatment protocols. One such protocol, entitled dose-adjusted EPOCH-R, utilizes two major new strategies. First, the treatment approach utilizes continuous infusion of chemotherapy over four days, instead of being administered over minutes or hours. Secondly, the doses of some medications involved are increased or decreased based on how the drugs affect the subject's ability to produce blood cells, which is used as a measure of how rapidly the body is processing drugs.

Using this approach in adults, researchers have shown improved cure rates in these cancers. Additionally, the harmful effects experienced by patients has been mild, with mucositis, severe infections, and tumor lysis syndrome occurring rarely. However, this new dosing method has never been used in children, and the effectiveness and side effects of this new method are unknown in children.

The purpose of this study is to look at the safety of dose-adjusted EPOCH-R in the treatment of children with mature B-cell cancers, and to see if we can maintain cure rates (as has been shown in adults). This study represents the first trial of dose-adjusted EPOCH-R in children.

DETAILED DESCRIPTION:
The subject will need to have a variety of tests, exams, or procedures to find out if s/he can be on the study.

The subject will also require placement of a catheter that stays in the vein for safe administration of chemotherapy drugs.

During the study...

If all of the tests that have been done show that s/he can participate and s/he chooses to participate, treatment cycles will begin.

A cycle equals three weeks. The subject will have a minimum of 6 cycles of treatment, possibly 8. The cancer drugs s/he will receive are etoposide, vincristine, doxorubicin, cyclophosphamide, prednisone, and rituximab with each cycle. The amount of the drugs will be determined by the subject's weight at first, and some of the drugs will be adjusted up or down for later cycles.

Rituximab will be given on Day 1 prior to continuous infusion drugs.

After 4 cycles, the subject will have imaging scans again to see how the cancer responded to treatment. If the cancer responds completely after 4 cycles, s/he will get 2 more cycles (6 cycles total). If the cancer partially responds, s/he will get 4 more cycles (8 total cycles).

If the subject has cancer in the Central Nervous System, s/he will receive a drug called methotrexate. If s/he does not have cancer in the CNS, s/he will get methotrexate to try to prevent CNS cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient with newly diagnosed, histologically confirmed, diffuse large B-cell lymphoma, or primary mediastinal B-cell lymphoma; or patient has post-transplant lymphoproliferative disorder regardless of when diagnosed.

Exclusion Criteria:

* Patient has received previous chemotherapy or radiation therapy in the three months prior to therapy, except for empiric initial intrathecal administration at diagnosis
* Patient who has received any prior anthracyclines.
* Patient with symptomatic cardiac failure unrelieved by medical therapy or evidence of significant cardiac dysfunction by echocardiogram (shortening fraction <28%) NOT due to mediastinal mass.
* Patient with severe renal disease (i.e. creatinine greater than 3 times normal for age; creatinine clearance less than 50 ml/min/1.73m2).
* Patient with severe hepatic disease (direct bilirubin greater than 3 mg/dl or AST greater than 500 IU/L).
* Patient with a Karnofsky performance score <50% or Lansky score <50%.
* Patient has been documented HIV positive and is unwilling/unable to stop antiretroviral therapy
* Female patient who is pregnant or breastfeeding.
* Patient is of reproductive potential and is not willing to use an acceptable method of birth control
* Patient has group classification A at diagnosis (completely resected stage I or completely resected stage II abdominal lesions)
* Patient has group classification B stage I or II disease with normal LDH level AND tumor mass less than 7 cm
* Patient has primary CNS lymphoma (lymphoma limited to the craniospinal axis without systemic involvement)
* Patient has Burkitt lymphoma or leukemia

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2013-01; Primary Completion 2016-08-26 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Measure and assess adverse events | 1 year
  To evaluate the safety and feasibility of dose-adjusted EPOCH-R in the treatment of use in children and young adults with mature B-cell malignancies, including, DLBCL, and PMBCL, as well as in patients with post-transplant lymphoproliferative disorder (PTLD).

SECONDARY OUTCOMES:
Measure and assess immune function | 1 year
  Blood will be taken to identify tumor and plasma biomarkers and mutations in patients with mature B-cell malignancies (DLBCL, PMBCL, and PTLD) that correlate with disease response and outcome using this novel therapeutic approach.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Allen, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States